CLINICAL TRIAL: NCT02516332
Title: Exercise and Pharmacotherapy for Anxiety in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00064329
Record Dates: First submitted 2015-07-30; First posted 2015-08-05 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Anxiety; Cardiovascular Disease
MeSH Terms: conditions — Anxiety Disorders; Cardiovascular Diseases | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supervised Aerobic Exercise (Experimental): Patients will exercise three times per week, under medical supervision, at a level of 70-85% of their VO2peak as determined at the time of their baseline exercise stress test. Patients' exercise will consist of 10 minutes of gradual warm-up exercises followed by 35 minutes of continuous walking, biking, or jogging, and 5 minutes of cool down exercises for a total a 50 minutes per session. Patients will be instructed to monitor their radial pulses and will be checked at least three times per session to ensure that they are within their prescribed exercise training ranges.
  Interventions: Behavioral: Supervised Aerobic Exercise
- Lexapro (Experimental): Treatment in the medication will be supervised by a study psychiatrist. Drug dispensing will be done by licensed pharmacists at the Duke Investigational Pharmacy Service. The investigators will use the SSRI escitalopram (Lexapro), which has received FDA approval for the treatment of anxiety, in 5 mg capsules. Medication will be dispensed as capsules of escitalopram in individually coded bottles. Medication adherence will be assessed using pill count at each study visit. Patients will visit face-to-face with a study psychiatrist at week 0 (baseline), week 1, week 2, week 4, week 8, and week 12 with phone encounters at weeks 3 and 6. The psychiatrist will make all medication adjustments based primarily upon Spielberger Anxiety Scores. Depending on symptoms, daily escitalopram doses will be titrated to 10 mg after week 2 and to 15 mg or placebo equivalent at week 3 if patients show no change or only minimal improvement.
  Interventions: Drug: Lexapro
- Placebo (Placebo Comparator): Treatment in the medication and placebo pill arms will be supervised by a study psychiatrist. Drug dispensing will be done by licensed pharmacists at the Duke Investigational Pharmacy Service, who have extensive experience in clinical trials. Medication will be taken once daily in the morning but can be switched to once daily in the evening if deemed necessary. Placebo medication administration will follow the same protocol as outlined for Lexapro.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lexapro
  Arms: Lexapro
Drug: Placebo
  Arms: Placebo
Behavioral: Supervised Aerobic Exercise
  Arms: Supervised Aerobic Exercise

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death in the United States; more than 600,000 Americans suffer a fatal cardiac event each year. Traditional CHD risk factors such as high blood pressure, smoking, and elevated cholesterol do not fully account for the timing and occurrence of CHD events and individuals with elevated levels of anxiety appear to have a greater risk of cardiovascular events. The present study will examine the impact of aerobic exercise and Lexapro in the treatment of anxiety and cardiovascular biomarkers among individuals with CHD.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of death in the United States; more than 600,000 Americans suffer a fatal cardiac event each year. Traditional CHD risk factors such as high blood pressure, smoking, and elevated cholesterol do not fully account for the timing and occurrence of CHD events. The term "cardiovascular vulnerable patient" has been used to describe patients susceptible to acute coronary events based upon plaque, blood, or myocardial characteristics. Psychosocial factors also have been shown to be associated with increased adverse health outcomes and increased cardiovascular vulnerability. For example, clinical depression and elevated depressive symptoms are associated with increased morbidity and mortality, and as a result, the American Heart Association has recommended that clinicians should routinely assess depression in CHD patients. Although much research and clinical recommendations have focused on depression, the significance of anxiety has been largely ignored, despite the fact that anxiety disorders are as prevalent as depression in the general population and are associated with similar levels of disability.

Despite the prevalence and prognostic significance of anxiety in CHD populations, there have been few randomized clinical trials (RCTs) specifically targeting anxious CHD patients. Anxiolytic medications, including selective serotonin reuptake inhibitors (SSRIs), have been shown to be effective in treating anxiety. SSRIs have been evaluated for the treatment of clinical depression in cardiac patients, with equivocal results. Surprisingly, to our knowledge, there have been no RCTs examining the efficacy of medications for treating anxiety in CHD patients. Moreover, because many cardiac patients are reluctant to take additional medications and psychotropic medications may not be effective for everyone or may produce unwanted side effects, there continue to be a need to identify alternative approaches for treating anxiety in cardiac patients. The investigators believe that exercise may be one such approach.

The purpose of this study is to evaluate the following hypotheses in a population of CHD patients with elevated symptoms of anxiety. The present study will examine the impact of a 3-month intervention of either exercise, Lexapro, or placebo on anxiety symptoms and CHD biomarkers among individuals with cardiac disease and elevated anxiety. The investigators hypothesize that: (1) Both exercise training and medication will reduce anxiety symptoms to a greater extent than placebo; (2) Exercise training will improve CHD biomarkers of risk including autonomic regulation, vascular endothelial function, and inflammation more than either medication or placebo; and (3) Improvements in CHD biomarkers will be mediated by reductions in symptoms of anxiety. The investigators also will explore potential moderators of treatment (e.g., anxiety diagnoses, CHD severity) as well as the longer-term benefits of treatment by documenting medical events and health care costs over a follow-up period of up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with documented CHD (i.e., a prior MI, coronary revascularization procedure, or >70% stenosis in at least one coronary artery)
* Age > 39 years
* Patients also will have an anxiety symptom severity score of at least 8 on the Hospital Anxiety and Depression-Anxiety scale (HADS-A) or a DSM-5 diagnosis of an Anxiety Disorder, such as General Anxiety, Social Anxiety, or Panic Disorder.

The study team plans to actively recruit women and minorities, with at least 50% women and 25% minorities.

Exclusion Criteria:

* An MI or coronary revascularization procedure (i.e., CABG or percutaneous coronary intervention) within the last 3 months
* Unstable angina
* Severe left ventricular dysfunction (ejection fraction <30%) or decompensated heart failure
* Unrevascularized left main coronary artery stenosis >50%
* Complete Pacemaker dependence
* Resting BP >200/120 mm Hg
* Conditions that would preclude randomization to either the drug (e.g., prolonged QT interval, known allergy to or intolerance of escitalopram) or exercise (e.g., musculoskeletal problems or abnormal cardiac response to exercise)
* Patients with a primary psychiatric diagnosis other than Anxiety Disorder will be excluded, including patients with PTSD, OCD, or any of the following DSM-5 diagnoses:

  1. Dementia, delirium;
  2. Schizophrenia, Schizoaffective, or other psychotic disorder;
  3. Psychotic features including any delusions or hallucinations; or
  4. Current alcohol or other substance abuse disorder.
* Similarly, patients who pose an acute suicide or homicide risk or who, during the course of the study, would likely require treatment with additional psychopharmacologic agents will not be enrolled.
* Patients will also be excluded if they are taking other medications that would preclude assignment to either drug or exercise conditions (e.g., clonidine, dicumarol, anticonvulsants, and MAO inhibitors) or are taking herbal supplements with purported mood effects (e.g., St. John's Wort, valerian, ginkgo).
* Patients already engaged in regular exercise (at least 30 minutes >1x/week) will not be enrolled.
* Finally, pregnant women will be excluded from participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-12; Primary Completion 2020-05-01 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Blumenthal JA, Smith PJ, Jiang W, Hinderliter A, Watkins LL, Hoffman BM, Kraus WE, Liao L, Davidson J, Sherwood A. Effect of Exercise, Escitalopram, or Placebo on Anxiety in Patients With Coronary Heart Disease: The Understanding the Benefits of Exercise and Escitalopram in Anxious Patients With Coronary Heart Disease (UNWIND) Randomized Clinical Trial. JAMA Psychiatry. 2021 Nov 1;78(11):1270-1278. doi: 10.1001/jamapsychiatry.2021.2236. PMID 34406354
- [Derived] Blumenthal JA, Feger BJ, Smith PJ, Watkins LL, Jiang W, Davidson J, Hoffman BM, Ashworth M, Mabe SK, Babyak MA, Kraus WE, Hinderliter A, Sherwood A. Treatment of anxiety in patients with coronary heart disease: Rationale and design of the UNderstanding the benefits of exercise and escitalopram in anxious patients WIth coroNary heart Disease (UNWIND) randomized clinical trial. Am Heart J. 2016 Jun;176:53-62. doi: 10.1016/j.ahj.2016.03.003. Epub 2016 Mar 12. PMID 27264220

RESULTS

PARTICIPANT FLOW:
Groups:
- Supervised Aerobic Exercise: Patients will exercise three times per week, under medical supervision, at a level of 70-85% of their VO2peak as determined at the time of their baseline exercise stress test. Patients' exercise will consist of 10 minutes of gradual warm-up exercises followed by 35 minutes of continuous walking, biking, or jogging, and 5 minutes of cool down exercises for a total a 50 minutes per session. Patients will be instructed to monitor their radial pulses and will be checked at least three times per session to ensure that they are within their prescribed exercise training ranges.
  Supervised Aerobic Exercise
- Lexapro: Treatment in the medication will be supervised by a study psychiatrist. Drug dispensing will be done by licensed pharmacists at the Duke Investigational Pharmacy Service. The investigators will use the SSRI escitalopram (Lexapro), which has received FDA approval for the treatment of anxiety, in 5 mg capsules. Medication will be dispensed as capsules of escitalopram in individually coded bottles. Medication adherence will be assessed using pill count at each study visit. Patients will visit face-to-face with a study psychiatrist at week 0 (baseline), week 1, week 2, week 4, week 8, and week 12 with phone encounters at weeks 3 and 6. The psychiatrist will make all medication adjustments based primarily upon Spielberger Anxiety Scores. Depending on symptoms, daily escitalopram doses will be titrated to 10 mg after week 2 and to 15 mg or placebo equivalent at week 3 if patients show no change or only minimal improvement.
  Lexapro
- Placebo: Treatment in the medication and placebo pill arms will be supervised by a study psychiatrist. Drug dispensing will be done by licensed pharmacists at the Duke Investigational Pharmacy Service, who have extensive experience in clinical trials. Medication will be taken once daily in the morning but can be switched to once daily in the evening if deemed necessary. Placebo medication administration will follow the same protocol as outlined for Lexapro.
  Placebo
Period: Overall Study
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Started | 52 | 53 | 23
Completed | 50 | 52 | 21
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo | Total
Number analyzed (Participants) | 52 | 53 | 23 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.1) | 63.9 (8.6) | 65.2 (10.8) | 64.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 6 | 37
  Male | 35 | 39 | 17 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 51 | 53 | 23 | 127
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 5
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 12 | 5 | 25
  White | 40 | 36 | 18 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 53 | 23 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change in Hospital Anxiety and Depression Scale (HADS), Anxiety
Description: The Hospital Anxiety and Depression Scale, Anxiety, is a 7-item subscale with scores ranging from 0-21, with higher scores indicating more anxiety.
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
score on a scale | -3.9 [-4.6 to -3.2] | -5.7 [-6.4 to -5.0] | -3.5 [-4.6 to -2.5]
Statistical Analysis 1: Comparison: Supervised Aerobic Exercise vs Lexapro vs Placebo; Test type: Other; p = 0.038, ANCOVA
Statistical Analysis 2: Comparison: Supervised Aerobic Exercise vs Lexapro vs Placebo; Test type: Other; p = 0.002, ANCOVA

2. Secondary Outcome: Change in Heart Rate Variability, SDNN (Msec)
Description: To quantify heart rate variability (HRV), an electrocardiogram was recorded for 24-hours using the 3-channel DigiTrak XT Holter recorder (Philips Healthcare, Andover, Massachusetts). Electrocardiographic data were downloaded and edited using the Philips Zymed Holter analysis software (2010 Plus/1810 series) and HRV was estimated from the standard deviation of the normal-to-normal R-R intervals (SDNN).
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
msec | -0.3 [-22.5 to 22.0] | -8.7 [-31.4 to 13.9] | -1.1 [-37.1 to 35.0]

3. Secondary Outcome: Change in Baroreflex Sensitivity, ms/mm Hg
Description: To assess baroreflex sensitivity (BRS), beat-by-beat systolic blood pressure (SBP) and heart rate (HR) were collected using the Nexfin noninvasive BP monitor (Bmeye, Amsterdam, Netherlands). BRS was estimated from the magnitude of the transfer function relating R-R interval oscillations to SBP oscillations across the 0.07 to 0.1299 Hz, or low frequency band.
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: ms/mm Hg
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
ms/mm Hg | 1.2 [-7.0 to 9.4] | 1.3 [-4.9 to 7.4] | 1.5 [-10.6 to 13.6]

4. Secondary Outcome: Change in Vascular Endothelial Function, Percentage of Dilation
Description: Endothelial function, assessed by Flow-Mediated Dilation (FMD), was determined from longitudinal B-mode ultrasound images of the brachial artery. Images were obtained using an Acuson (Mountain View, California) Aspen ultrasound platform with an 11-MHz linear-array transducer after 10 min of supine relaxation and during reactive hyperemia, induced by the inflation of a forearm pneumatic occlusion cuff to suprasystolic pressure (about 200 mm Hg) and subsequent deflation after 5 min. FMD was defined as the maximum percentage change in arterial diameter relative to resting baseline from 10 to 120 s after deflation of the occlusion cuff.
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of dilation
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
percentage of dilation | 0.7 [-0.2 to 1.5] | 0.5 [-0.4 to 1.3] | 0.5 [-0.8 to 1.8]

5. Secondary Outcome: Change in Inflammation (C-Reactive Protein, ug/ml)
Description: High-sensitivity C-reactive protein was quantified by ELISA (LabCorp). Values >10 mg/L were truncated at 10 to account for acute inflammatory processes that may have skewed the distribution of this blood marker.
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
ug/ml | -0.2 [-3.0 to 2.5] | 0.1 [-2.0 to 2.2] | -0.3 [-4.0 to 3.4]

6. Secondary Outcome: Change in Urinary Catecholamines (Epinephrine and Norepinephrine, Unit-weighted Z-score)
Description: Urinary catecholamines, an index of sympathetic nervous system (SNS) activity, served as a biomarker of anxiety. Urinary concentrations of epinephrine (EPI) and norepinephrine (NE) were determined by high-pressure liquid chromatography (HPLC) with electrochemical detection (LabCorp). A composite 24-hr catecholamines z-score is presented. The z-score is the raw score minus the population mean, divided by the population standard deviation. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
z-score | 0.05 [-0.2 to 0.3] | -0.24 [-0.4 to 0.0] | 0.36 [0.0 to 0.7]
Statistical Analysis 1: Comparison: Supervised Aerobic Exercise vs Placebo; Test type: Other; p = 0.011, Regression, Linear
Statistical Analysis 2: Comparison: Supervised Aerobic Exercise vs Lexapro; Test type: Other; p = 0.036, Regression, Linear

7. Secondary Outcome: Change in Lipids - Total Cholesterol, LDL (Low-density Lipoprotein), and HDL (High-density Lipoprotein); mg/dL
Description: Lipids were obtained from fasting blood samples and assays were measured enzymatically (LabCorp).
Time Frame: Baseline, 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
Number analyzed (Participants) | 52 | 53 | 23
mg/dL
  Total Cholesterol | -28.2 [-67.3 to 10.8] | -15.3 [-50.6 to 20.0] | -31.6 [-90.2 to 27.1]
  LDL | -18.6 [-46.3 to 9.2] | -9.8 [-33.5 to 13.9] | -19.3 [-59.9 to 21.4]
  HDL | 6.3 [-4.4 to 16.9] | 3.4 [-5.5 to 12.4] | 7.2 [-8.3 to 22.7]

8. Other Pre Specified Outcome: Change in Hospital Anxiety and Depression Scale, Total Score
Time Frame: 9 months, 15 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 3 months
Groups:
- Supervised Aerobic Exercise: Patients will exercise three times per week, under medical supervision, at a level of 70-85% of their VO2peak as determined at the time of their baseline exercise stress test. Patients' exercise will consist of 10 minutes of gradual warm-up exercises followed by 35 minutes of continuous walking, biking, or jogging, and 5 minutes of cool down exercises for a total a 50 minutes per session. Patients will be instructed to monitor their radial pulses and will be checked at least three times per session to ensure that they are within their prescribed exercise training ranges.
  Supervised Aerboic Exercise
Arm/Group | Supervised Aerobic Exercise | Lexapro | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/23
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT02516332/Prot_SAP_000.pdf